CLINICAL TRIAL: NCT06856135
Title: Expanded Access Program for United States of America: Vedolizumab Intravenous for the Treatment of Pediatric Patients With Moderate to Severe Ulcerative Colitis or Crohn's Disease
Brief Title: Expanded Access to Vedolizumab for Children and Teenagers With Ulcerative Colitis or Crohn's Disease in the USA
Status: Available | Type: Expanded Access
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vedolizumab 4072
Record Dates: First submitted 2025-02-25; First posted 2025-03-04 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: Drug Therapy
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Vedolizumab IV — Participants will continue to receive vedolizumab IV at the same dose administered at the end of Trial Vedolizumab-2005 (NCT03196427), at a frequency of every 8 weeks.
  • Other Names:
  * MLN0002
  * ENTYVIO
  * KYNTELES

SUMMARY:
The expanded access program (EAP) allows people to gain access to an unlicensed treatment on compassionate grounds. This EAP provides children and teenagers with Ulcerative Colitis (UC) or Crohn's Disease (CD) who completed the Vedolizumab-2005 clinical study in the United States (US) with continued access to Vedolizumab Intravenous (IV) which is given as infusion into a vein (intravenously IV) until it becomes commercially available in the US. To be able to participate in this EAP, children and teenagers must still benefit from the treatment with Vedolizumab IV. According to the participant's treating healthcare professional (HCP): there are no comparable and satisfactory alternative treatment options in the local market, or the participant would be negatively affected without continued access to vedolizumab IV.

ELIGIBILITY:
Inclusion Criteria:

1. The participant has UC or CD and is of age less than (<) 18 years at the time of final treatment completion of Vedolizumab-2005.
2. The participant is demonstrating continued clinical benefit from vedolizumab IV for the treatment of UC or CD that outweighs possible risks.
3. The participant, participant's legally authorized representative, or adult caregiver is informed of the nature of this expanded access program and has provided signed and dated written informed consent and/or pediatric assent.
4. The participant does not have any condition, including laboratory test result, that in the opinion of the investigator may compromise the participant's safety.
5. The participant does not have a known hypersensitivity to vedolizumab or its components.
6. According to the participant's treating healthcare professional (HCP): there are no comparable and satisfactory alternative treatment options in the local market, or the participant would be negatively affected without continued access to vedolizumab IV.
7. Female participants of childbearing potential only:

   * The participant has agreed to be abstinent or agreed to comply with the applicable contraceptive requirements of this protocol for the duration of the expanded access program and for 18 weeks after completion of the last dose of vedolizumab.
   * The participant is not pregnant or breastfeeding.
   * The participant will not donate ova during the course of the program and for 18 weeks after the last dose of vedolizumab.
8. Male participants only:

   * The participant has agreed to comply with the applicable contraceptive requirements of this protocol for the duration of the expanded access program and for 18 weeks after the last dose of vedolizumab.
   * The participant has agreed to not donate sperm during the course of the program and for 18 weeks after the last dose of vedolizumab.

Exclusion Criteria:

-No specific exclusion criteria.

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- United States (3):
  - University of California San Francisco, San Francisco, California
  - Children's Center for Digestive Healthcare, Atlanta, Georgia
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language. — https://clinicaltrials.takeda.com/study-detail/9a18ff51d4d2479a??page=1&idFilter=Vedolizumab+4072